CLINICAL TRIAL: NCT03543293
Title: Fast and Accurate Diagnosis of an Oval or Round Window Perilymphatic Fistula on CT and MRI, Without Injection, on 101 Patients With Surgical Confirmation
Brief Title: Imaging Perilymphatic Fistulas After Barotrauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6807
Record Dates: First submitted 2018-02-26; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-02

CONDITIONS: Perilymphatic Fistulas
Keywords: perilymphatic fistulas; magnetic resonance imaging (MRI); surgery; round window; vertigo; tinnitus; cophosis
MeSH Terms: conditions — Vertigo; Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to validate the CT / MRI combination of non-injected rock for the rapid positive diagnosis of perilymphatic fistulas.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Clinical suspicion of perilymphatic fistula
* Patient having undergone a rock scan or MRI of the middle ear at the Strasbourg University Hospital with surgical confirmation of the diagnosis (or reversal)

Exclusion Criteria:

- Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having undergone a rock scan or MRI of the middle ear at the Strasbourg University Hospital with surgical confirmation of the diagnosis (or reversal)
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of perilymphatic fistula | 1 hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francis VEILLON, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No